CLINICAL TRIAL: NCT07363408
Title: A Phase I Clinical Trial of Ivonescimab and ADG126, Alone, and in Combination With 5-FU/LV or FOLFIRI in MSS Advanced/Metastatic Colorectal Cancer
Brief Title: Ivonescimab and ADG126, Alone, and in Combination With Leucovorin and Fluorouracil or FOLFIRI Regimen for the Treatment of Microsatellite Stable Advanced/Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25512; NCI-2025-09719 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25512 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Microsatellite Stable Colorectal Carcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Specimen Handling; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (muzastotug, ivonescimab) (Experimental): Patients receive muzastotug IV over 60-90 minutes on day 1 of each cycle and ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, and collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ivonescimab; Procedure: Magnetic Resonance Imaging; Biological: Muzastotug
- Arm B (muzastotug, ivonescimab, leucovorin, fluorouracil) (Experimental): Patients receive muzastotug IV over 60-90 minutes on day 1 of each cycle, ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle, leucovorin IV over 2 hours on days 1, 15, and 29 of each cycle, and fluorouracil IV continuously over 46 hours on days 1, 15, and 29 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, and collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Biological: Ivonescimab; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Biological: Muzastotug
- Arm C (muzastotug, ivonescimab, FOLFIRI) (Experimental): Patients receive muzastotug IV over 60-90 minutes on day 1 of each cycle, ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle, leucovorin IV over 2 hours on days 1, 15, and 29 of each cycle, fluorouracil IV continuously over 46 hours on days 1, 15, and 29 of each cycle, and irinotecan IV over 90 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, and collection of blood samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Irinotecan; Biological: Ivonescimab; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Biological: Muzastotug

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm B (muzastotug, ivonescimab, leucovorin, fluorouracil); Arm C (muzastotug, ivonescimab, FOLFIRI)
Drug: Irinotecan — Given IV
  Arms: Arm C (muzastotug, ivonescimab, FOLFIRI)
Biological: Ivonescimab — Given IV
  Other Names: AK 112; AK-112; AK112; Anti-PD-1/Anti-VEGF Bispecific Antibody AK112; Anti-PD-1/VEGF Bispecific Antibody AK112; PD-1/VEGF Bispecific Antibody AK112; SMT 112; SMT-112; SMT112
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm B (muzastotug, ivonescimab, leucovorin, fluorouracil); Arm C (muzastotug, ivonescimab, FOLFIRI)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Muzastotug — Given IV
  Other Names: ADG 126; ADG-126; ADG126; Anti-CTLA-4 Monoclonal Antibody ADG126; Anti-CTLA-4 SAFEbody ADG126

SUMMARY:
This phase I trial studies the safety, side effects, and best dose of ADG126, in combination with ivonescimab alone, in combination with ivonescimab, leucovorin, and fluorouracil, or in combination with ivonescimab and leucovorin, fluorouracil, and irinotecan (FOLFIRI regimen) in treating patients with microsatellite stable (MSS) colorectal cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or has spread from where it first started (primary site) to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as ivonescimab and ADG126, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ivonescimab may also stop or slow the cancer by blocking the growth of new blood vessels necessary for tumor growth. Leucovorin calcium is a type of drug called a folic acid analog, which means it is similar to the vitamin folic acid. It is used in combination with certain chemotherapy drugs to enhance their ability to kill tumor cells or to lessen their harmful side effects. Fluorouracil is a type of chemotherapy called an antimetabolite, which is a drug that mimics a natural chemical and prevents its use in cells. It interferes with the production of a key component of deoxyribonucleic acid (DNA), which prevents the DNA from copying itself. This causes tumor cells and other rapidly dividing cells to die. Fluorouracil also gets incorporated into ribonucleic acid (RNA) and DNA, disrupting critical cell functions. Irinotecan is in a class of antineoplastic medications called topoisomerase I inhibitors. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Giving ADG126 with ivonescimab, with or without leucovorin and fluorouracil or FOLFIRI regimen, may be safe in treating patients with MSS advanced/metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended phase II dose of muzastotug (ADG126) and ivonescimab (Arm A) in advanced/metastatic MSS colorectal cancer without liver metastatic disease.

II. Determine the recommended phase II dose of ADG126 and ivonescimab with fluorouracil (5-FU)/leucovorin (LV) (Arm B) in advanced/metastatic MSS colorectal cancer.

III. Determine the recommended phase II dose of ADG126 and ivonescimab with leucovorin, fluorouracil, and irinotecan (FOLFIRI) (Arm C) in advanced/metastatic MSS colorectal cancer.

SECONDARY OBJECTIVES:

I. Describe the safety of giving ADG126 with ivonescimab, and in combination with 5-FU/LV, and in combination with FOLFIRI in MSS advanced/metastatic colorectal cancer.

II. Describe the overall response rate (ORR) as evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for the three treatment arms individually.

III. Describe the duration of response (DoR), progression free survival (PFS), and overall survival (OS) of each of the three treatment arms.

IV. Assess ADG126 pharmacokinetics (PK) through sparse sampling at different doses of ADG126 on study and in combination with ivonescimab, 5-FU/LV, or FOLFIRI.

EXPLORATORY OBJECTIVE:

I. Explore the dynamics of immune cells in relation to clinical outcome by treatment arm, which include the data from immunophenotyping, cytokine analysis and ribonucleic acid (RNA) sequencing of peripheral blood and buffy coat at baseline, 4 weeks, and 8 weeks, and every subsequent 8 weeks until progression.

OUTLINE: This is a dose-escalation study of muzastotug in combination with ivonescimab, leucovorin, fluorouracil, and irinotecan. Patients are assigned to 1 of 3 arms.

ARM A: Patients receive muzastotug intravenously (IV) over 60-90 minutes on day 1 of each cycle and ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI), and collection of blood samples throughout the study.

ARM B: Patients receive muzastotug IV over 60-90 minutes on day 1 of each cycle, ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle, leucovorin IV over 2 hours on days 1, 15, and 29 of each cycle, and fluorouracil IV continuously over 46 hours on days 1, 15, and 29 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, and collection of blood samples throughout the study.

ARM C: Patients receive muzastotug IV over 60-90 minutes on day 1 of each cycle, ivonescimab IV over 60 minutes on days 1, 15, and 29 of each cycle, leucovorin IV over 2 hours on days 1, 15, and 29 of each cycle, fluorouracil IV continuously over 46 hours on days 1, 15, and 29 of each cycle, and irinotecan IV over 90 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI, and collection of blood samples throughout the study.

After completion of study treatment, patients are followed for 30 days, every 3 months until disease progression (if applicable) for 2 years and/or after disease progression periodically for survival.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Agreement to blood collection for correlative analysis at baseline, 4 weeks, and 8 weeks, and then every subsequent 8 weeks
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Histologically confirmed advanced/metastatic MSS colorectal cancer. MSS status must have been confirmed by a Clinical Laboratory Improvement Amendments (CLIA) certified assay
* Measurable disease by RECIST 1.1
* Fully recovered from the acute, clinically significant, toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* ARM A ONLY: Patients should not have evidence of hepatic metastatic disease
* ARM A ONLY: Patients should have progressed following irinotecan, oxaliplatin, fluoropyrimidine, and an anti-EGFR if clinically indicated
* ARM B ONLY: Patient is eligible for maintenance 5-FU/LV or 5-FU/LV bevacizumab
* ARM B ONLY: No history of significant toxicity to 5-FU/LV that required dose reduction in infusional 5-FU dosing
* ARM C ONLY: Patient is eligible for FOLFIRI chemotherapy
* ARM C ONLY: No history of significant toxicity to 5-FU/LV or irinotecan that required dose reduction in infusional 5-FU dosing or irinotecan
* ARM C ONLY: No prior progression on prior irinotecan and no prior dose reduction on irinotecan due to toxicity
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L

  * NOTE: no blood transfusions or growth factor therapy used within 7 days of the screening complete blood count (CBC)
* Platelets ≥ 100 × 10^9/L

  * NOTE: no blood transfusions or growth factor therapy used within 7 days of the screening CBC
* Hemoglobin ≥ 9.0 g/dL

  * NOTE: no blood transfusions or growth factor therapy used within 7 days of the screening CBC
* Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); For patients with liver metastases or confirmed/suspected Gilbert syndrome, TBIL ≤ 3 × ULN
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN; For patients with liver metastases ≤ 5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN; For patients with liver metastases ≤ 5 x ULN
* Creatinine clearance of ≥ 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥ 30 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (adjustment by body surface area [BSA] is not required for eGFR; eGFR can be determined using the calculator from the National Kidney Foundation website [www.kidney.org])
* International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN (unless abnormalities are unrelated to coagulopathy). This applies only to patients who are not on therapeutic anti-coagulation. Patients receiving therapeutic anti-coagulation should be on a stable dose
* Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g
* For patients with KNOWN history of HIV, hepatitis C virus (HCV) and/or hepatitis B virus (HBV) seropositivity only, nucleic acid quantitation for their virus must be performed.

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load and a cd4 > 400 are eligible for this trial.
  * Patients with known active hepatitis B are required to have hepatitis B DNA < 200 IU/ml by polymerase chain reaction (PCR) and on appropriate anti-viral therapy with acceptable tolerability for one month prior to randomization.
  * All patients with known active hepatitis C (hepatitis C virus [HCV] antibody positive with HCV RNA levels above the lower limit of detection) are excluded
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 6 months after the last dose of study drug. Unsterilized male patients having sex with a female partner of childbearing potential, or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 6 months after the last dose of study drug. Male patients with female partners of childbearing potential must have the female partner agree to use at least 1 form of highly effective contraception for the duration of the treatment period until 6 months after the last dose of study drug

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Major surgical procedures or serious trauma within 4 weeks prior to study entry, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to study entry
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days or five half-lives (whichever is shorter for non-radiation therapy) prior to day 1 of protocol therapy
* Strong CYP3A4 inducers/ inhibitors within 14 days prior to day 1 of protocol therapy (Arm C only)
* UGT1A1 inhibitors within 14 days prior to day 1 of protocol therapy (Arm C only)
* Any other anti-cancer therapy is prohibited, including but not limited to antibody-based therapy, retinoids, nitrosourea therapy, mitomycin C, small molecule tyrosine kinase inhibitors, proprietary Chinese medicines with anti-cancer activity, or radiotherapy
* Herbal medications must be cleared by the principal investigator (PI)
* Prior exposure to PD-1 or PD-L1 or CTLA-4 targeting agents
* History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to study entry, including but not limited to:

  * Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots) Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed
  * Nasal bleeding/epistaxis (bloody nasal discharge is allowed)
  * Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to study entry is not allowed. The use of full-dose anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits according to the medical standard of the enrolling institution or with the use of factor Xa inhibitors
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
* Active autoimmune or lung disease requiring systemic therapy (eg, with disease modifying drugs, prednisone > 10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to study entry, however the following will be allowed:

  * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
  * Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted
* History of major diseases before study entry, specifically:

  * Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or unstable vascular disease (eg, aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to study entry, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
  * History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months before study entry
  * History of any grade arterial thromboembolic event, grade 3 and above venous thromboembolic event, as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to study entry
  * Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks before study entry
  * History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to study entry
* Imaging during the screening period shows that the patient has:

  * Radiologically documented evidence of major blood vessel invasion or fistula
* Symptomatic central nervous system (CNS) metastases, CNS metastases with hemorrhagic features, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to study entry, potential need for CNS radiation within the first cycle, or leptomeningeal disease. Note: Patients must have stopped corticosteroids or be on physiologic corticosteroid replacement therapy (prednisone ≤ 10 mg daily or equivalent)
* Live vaccine or live attenuated vaccine within 4 weeks prior to planned study entry, or if scheduled to receive a live vaccine or live attenuated vaccine during the study period. Inactivated vaccines are permitted
* Severe infection within 4 weeks prior to study entry, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection (as determined by the investigator) requiring systemic anti-infective therapy within 2 weeks prior to study entry, (excluding antiviral therapy for hepatitis B or C)
* Has pre-existing peripheral neuropathy that is ≥ grade 2 by CTCAE version 5.0
* Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic or required paracentesis in the last 4 weeks prior to enrollment
* History of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease
* Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Current use of systemic corticosteroids (>10 mg daily prednisone or equivalent)
* High risk for bowel perforation such as obstructive gastrointestinal (GI) findings on imaging or symptoms suggesting bowel obstruction (post-prandial cramping, nausea, or vomiting)
* Presence of an enteric stent
* Open non-healing wounds
* History of bowel perforation unless related to the primary tumor and unless the tumor was resected or the patient has been diverted proximal to the tumor
* Known allergy to any component of any study drug; known history of severe hypersensitivity to other monoclonal antibodies; history of allergic reactions attributed to compounds of similar chemical or biologic composition to any study agent
* History or current evidence of any condition (medical [including adverse events from prior anticancer therapy, disorders secondary to tumor], surgical or psychiatric [including substance abuse]), or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, might lead to higher medical risk and/or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Clinically significant uncontrolled illness
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient is breastfeeding or plans to breastfeed during the study
* Females only: Pregnant
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07-21 (Estimated); Primary Completion 2027-07-21 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Up to 6 weeks or 3 doses of ivonescimab, whichever is longer
  Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, by treatment arm. Descriptive statistics will be used for all safety, efficacy and immunogenicity parameters. Data will be summarized using descriptive statistics (number of subjects, mean, median, standard deviation, minimum, and maximum) for continuous variables and using frequencies and percentages for categorical variables. Differences among groups will be tested using the Fisher's exact test and Kruskal-Wallis test for categorical and continuous variables, respectively.

SECONDARY OUTCOMES:
Treatment-related adverse event rates | Up to 30 days after completion of study treatment
  Will be assessed by NCI CTCAE version 5.0, delineated by grade and attribution, by treatment arm. Descriptive statistics will be used for all safety, efficacy and immunogenicity parameters. Data will be summarized using descriptive statistics (number of subjects, mean, median, standard deviation, minimum, and maximum) for continuous variables and using frequencies and percentages for categorical variables. Differences among groups will be tested using the Fisher's exact test and Kruskal-Wallis test for categorical and continuous variables, respectively.
Objective response rate | From the start of the study treatment and disease progression or death due to any cause prior to receiving another therapy, whichever occurs first, assessed up to 2 years after completion of study treatment
  Defined as rate of participants achieving confirmed complete response (CR) or partial response (PR), as assessed by the investigator using Response Evaluation Criteria in Solid Tumors 1.1. The point estimate and 95% confidence intervals will be provided using the Clopper-Pearson methods. Logistic regression modeling of responders (CR or PR) and non-responders will be used to estimate the level of association of treatment and objective response.
Duration of response | From the time when a response is experienced to progression or death, assessed up to 2 years after completion of study treatment
  Survival distributions will be estimated using the Kaplan-Meier (KM) method. Survival curves will be compared between groups using the log-rank test. Median and landmark time-point estimates will be based on the KM estimates. The average hazard ratios (HR) will be estimated using a Cox proportional-hazards model. An assessment of the proportional-hazards assumption will be performed, and an assessment of the time-dependent HR will be done.
Progression-free survival | From the start of treatment to disease progression or death from any cause, whichever occurs first, assessed up to 2 years after completion of study treatment
  Survival distributions will be estimated using the KM method. Survival curves will be compared between groups using the log-rank test. Median and landmark time-point estimates will be based on the KM estimates. The average HR will be estimated using a Cox proportional-hazards model. An assessment of the proportional-hazards assumption will be performed, and an assessment of the time-dependent HR will be done.
Overall survival | From start of treatment to death due to any cause, assessed up to 2 years after completion of study treatment
  Survival distributions will be estimated using the KM method. Survival curves will be compared between groups using the log-rank test. Median and landmark time-point estimates will be based on the KM estimates. The average HR will be estimated using a Cox proportional-hazards model. An assessment of the proportional-hazards assumption will be performed, and an assessment of the time-dependent HR will be done.
Plasma concentrations of cleaved and intact ADG126 | Up to 30 days after completion of study treatment
  Changes over time in the levels of biomarkers will be measured using Wilcoxon signed rank test and linear mixed effect model.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States